CLINICAL TRIAL: NCT00159523
Title: The Impact of Perinatal Daily Supplement of a Probiotic (Lactobacillus Rhamnosus GG), Given to Mothers, on Immunological Development, Atopic Sensitisation and Allergic Disease in Their Off-spring
Brief Title: Impact in Off-spring of Mothers After Perinatal Daily Intake of a Probiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Tine (Industry); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 097-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-08

CONDITIONS: Asthma; Dermatitis, Atopic; Rhinitis, Allergic, Perennial
Keywords: Prevention; Probiotics; Allergy; Hypersensitivity
MeSH Terms: conditions — Asthma; Dermatitis, Atopic; Rhinitis, Allergic, Perennial; Hypersensitivity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Other Names: Lactobacillus rhamnosus GG
  Arms: probiotic
Biological: placebo
  Arms: placebo

SUMMARY:
A probiotic (Lactobacillus rhamnosus GG) supplement to pregnant women the last four weeks of pregnancy and three months after birth is expected to give a 40% reduction in risk of atopic sensitisation and allergic disease at two years of age, compared to placebo.

DETAILED DESCRIPTION:
To investigate how probiotics given to pregnant women during the last 4 weeks of pregnancy and the first 4 months after birth influence the establishment and composition of the gut microflora in children from birth until two years of age.

At the same time to investigate the relationship between gut flora composition and the development of the immune system.

To investigate the relationship between supplement of probiotics to pregnant and breast-feeding women, the microbial composition of the gut flora in their children, the development of the childrens' immune system, and the prevalence of atopic sensitisation and atopic disease at two years of age.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women understanding Norwegian language and who has signed an informed consent form, can be included.
* Inclusion must take place before week 36 in the pregnancy.
* The woman must plan to breast-feed the first 4 months after birth.
* She must live in Trondheim.

Exclusion Criteria:

* Not being able to fill in the questionnaire in Norwegian language
* Lactose intolerance
* Consumption of probiotics earlier in the pregnancy.
* Intention to move from Trondheim in the next 25 months.
* Pregnant women in risk of eclampsia, or other serious disease that can influence beast-feeding or care for the child.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 416 (Actual)
Dates: Start 2003-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Atopic disease defined as atopic eczema, allergic rhino conjunctivitis or asthma at two years of age | 2 years

SECONDARY OUTCOMES:
Atopic sensitization | 2 years
Positive skin prick test (SPT), elevated total IgE and elevated specific IgE | 2 years
Intestinal microflora | 2 years
Intestinal colonisation with LGG. | 2 years
Oral cavity colonisation with LGG. | 2 years
Immunomarkers | 2 years
TGF in breastmilk | 2 years
Cytokine profile from activated PBMC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Katarina Cartfjord, Director, Study Director — Faculty of Medicine, NTNU
Locations (1):
- Dep of Public health and general Practice, Trondheim, Norway

REFERENCES:
- [Result] Dotterud CK, Storro O, Johnsen R, Oien T. Probiotics in pregnant women to prevent allergic disease: a randomized, double-blind trial. Br J Dermatol. 2010 Sep;163(3):616-23. doi: 10.1111/j.1365-2133.2010.09889.x. Epub 2010 Jun 9. PMID 20545688
- [Result] Simpson MR, Dotterud CK, Storro O, Johnsen R, Oien T. Perinatal probiotic supplementation in the prevention of allergy related disease: 6 year follow up of a randomised controlled trial. BMC Dermatol. 2015 Aug 1;15:13. doi: 10.1186/s12895-015-0030-1. PMID 26232126
- [Derived] Zakiudin DP, Ro ADB, Videm V, Oien T, Simpson MR. Systemic inflammatory proteins in offspring following maternal probiotic supplementation for atopic dermatitis prevention. Clin Mol Allergy. 2023 Jul 29;21(1):5. doi: 10.1186/s12948-023-00186-3. PMID 37516841
- [Derived] Schei K, Simpson MR, Avershina E, Rudi K, Oien T, Juliusson PB, Underhill D, Salamati S, Odegard RA. Early Gut Fungal and Bacterial Microbiota and Childhood Growth. Front Pediatr. 2020 Nov 9;8:572538. doi: 10.3389/fped.2020.572538. eCollection 2020. PMID 33240830
- [Derived] Schei K, Avershina E, Oien T, Rudi K, Follestad T, Salamati S, Odegard RA. Early gut mycobiota and mother-offspring transfer. Microbiome. 2017 Aug 24;5(1):107. doi: 10.1186/s40168-017-0319-x. PMID 28837002
- [Derived] Simpson MR, Ro AD, Grimstad O, Johnsen R, Storro O, Oien T. Atopic dermatitis prevention in children following maternal probiotic supplementation does not appear to be mediated by breast milk TSLP or TGF-beta. Clin Transl Allergy. 2016 Jul 22;6:27. doi: 10.1186/s13601-016-0119-6. eCollection 2016. PMID 27453775
- [Derived] Simpson MR, Brede G, Johansen J, Johnsen R, Storro O, Saetrom P, Oien T. Human Breast Milk miRNA, Maternal Probiotic Supplementation and Atopic Dermatitis in Offspring. PLoS One. 2015 Dec 14;10(12):e0143496. doi: 10.1371/journal.pone.0143496. eCollection 2015. PMID 26657066
- [Derived] Dotterud CK, Avershina E, Sekelja M, Simpson MR, Rudi K, Storro O, Johnsen R, Oien T. Does Maternal Perinatal Probiotic Supplementation Alter the Intestinal Microbiota of Mother and Child? J Pediatr Gastroenterol Nutr. 2015 Aug;61(2):200-7. doi: 10.1097/MPG.0000000000000781. PMID 25782657